CLINICAL TRIAL: NCT00012064
Title: Vaccine Biotherapy of Cancer: Tumor Cells and Dendritic Cells as Active Specific Immunotherapy of Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage IV or Recurrent Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068481; HOAG-VACCINE-MEL; NCI-V01-1646
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological/Vaccine (Experimental): Biological/Vaccine: therapeutic autologous dendritic cells.
  Apheresis procedure collects peripheral blood mononuclear cells (PBMC) for the production of dendritic cell, which are admixed with irradiated tumor cells from autologous tumor cell line for vaccine product.
  Interventions: Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells — Apheresis procedure collects peripheral blood mononuclear cells (PBMC) for the production of dendritic cell, which are admixed with irradiated tumor cells from autologous tumor cell line for vaccine product.

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have stage IV or recurrent melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of immunization with autologous in vitro-treated tumor cells and dendritic cells in combination with sargramostim (GM-CSF) in patients with stage IV or recurrent melanoma.
* Determine the frequency of conversion of delayed tumor hypersensitivity tests in patients treated with this regimen.
* Determine the progression-free and overall survival in patients treated with this regimen.
* Determine the objective tumor response rate in patients with measurable melanoma treated with this regimen.

OUTLINE: Patients are stratified according to presence of measurable disease at study initiation (yes vs no).

Patients undergo tumor cell harvest. Patients with multiple persistent sites of metastatic disease after harvest may receive systemic therapy (biologic therapy and/or chemotherapy) during tumor cell line expansion over approximately 4 months. The tumor cell line is expanded, irradiated, and treated with interferon gamma.

Patients undergo leukapheresis to collect peripheral blood mononuclear cells (PBMC) to obtain dendritic cells (DC). The PBMC are treated with sargramostim (GM-CSF) and interleukin-4 for 7 days to produce DC. The DC are then cultured with the treated tumor cells for 18 hours.

Patients undergo delayed tumor hypersensitivity tests intradermally 1 week prior to vaccination and again at week 4. Patients receive vaccine therapy comprising autologous treated tumor cells and dendritic cells suspended in GM-CSF subcutaneously weekly for 3 weeks. Vaccine therapy continues monthly for an additional 5 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 3 months for 4 years.

PROJECTED ACCRUAL: A total of 30-80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV or recurrent melanoma

  * Metastatic disease confirmed by MRI or CT scan
* Planned resection of tumor
* No active CNS metastases

  * Radiographically confirmed lack of CNS disease progression
  * No requirement for pharmacologic doses of corticosteroids

PATIENT CHARACTERISTICS:

Age:

* Over 16

Performance status:

* ECOG 0-2

Life expectancy:

* At least 4 months

Hematopoietic:

* Hematocrit greater than 25%
* Platelet count greater than 100,000/mm^3
* No ongoing transfusion requirements
* No active blood clotting or bleeding diathesis

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Albumin at least 3.0 g/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No underlying cardiac disease associated with known myocardial dysfunction
* No unstable angina related to atherosclerotic cardiovascular disease

Other:

* No other malignancy within the past 5 years except for carcinoma in situ, basal cell carcinoma, or localized squamous cell skin cancer
* No active, eminently life-threatening infection or medical condition
* Adequate venous access
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Other prior putative vaccines allowed
* Recovered from prior biologic therapy
* No other concurrent biologic therapy except epoetin alfa for patients with hematocrit less than 36%

Chemotherapy:

* At least 3 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent endocrine therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy (including whole brain radiotherapy) and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* Concurrent bisphosphonates allowed for patients with lytic bone metastases
* No concurrent digoxin or other medications designed to improve cardiac output
* No other concurrent investigational therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety of administration of irradiated autologous tumor cells that have been incubated in vitro with gamma interferon, and subsequently injected subcutaneously with autologous dendritic cells and GMCSF | treatment
To determine the frequency of conversion of delayed tumor hypersensitivity (DTH) tests with irradiated autologous tumor cells, in patients who received an autologous dendritic cell/tumor cell vaccine with GMCSF | treatment

SECONDARY OUTCOMES:
To determine the objective tumor response rate in patients with metastatic melanoma who still had measurable disease at the time vaccine treatment was given | follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Cancer Center at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Result] Dillman RO, Schiltz PM, Selvan R, et al.: Patient-specific cancer vaccine of cultured autologous tumor cells and autologous dendritic cells. [Abstract] J Immunother 24 (5): S5, 2001.